CLINICAL TRIAL: NCT07068685
Title: Pilot Testing Implementation of Suicide Risk Prediction Algorithms to Support Suicide Prevention in Primary Care
Brief Title: Pilot Testing Suicide Risk Prediction Algorithms in Primary Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019330; R34MH132829 (NIH)
Record Dates: First submitted 2025-07-02; First posted 2025-07-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Suicide Prevention; Suicide Risk | Patient
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Retrospective pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suicide risk monitoring (Experimental): Quality improvement intervention: 6 months following implementation of the suicide risk prediction algorithm in primary care to prompt extra mental health monitoring.
  Interventions: Other: Suicide risk prediction algorithm
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Suicide risk prediction algorithm — Use of a suicide risk prediction algorithm, developed by the Mental Health Research Network (MHRN), will be used to prompt additional mental health monitoring. Mental health monitoring will include asking patients about suicidal thoughts (via the ninth question of the Patient Health Questionnaire-9, PHQ-9), followed by suicide risk assessment (via use of a brief self-administered version of the Columbia Suicide Risk Severity Rating Scale, C-SSRS), followed by Safety Planning with a designated member of the primary care team.
  Other Names: suicide care clinical decision support
  Arms: Suicide risk monitoring

SUMMARY:
The goal of this pilot study is to learn whether the use of suicide risk prediction algorithms in primary care can help identify people who may benefit from extra mental health monitoring.

Specifically, this study aims to measure how use of the suicide risk prediction algorithm to prompt extra mental health monitoring among adult primary care patients impacts proportions of patients identified at risk of suicide and engaged in safety planning. Secondarily, we plan to measure proportions of patients identified at risk of suicide via mental health monitoring (irrespective of engagement in safety planning).

ELIGIBILITY:
Inclusion Criteria: Any type of adult primary care visit/encounter at Kaiser Permanente Washington (KPWA) between 3/5/25-10/5/25 (pre-period) and '10/6/25-4/5/26 (post-period or implementation period).

Exclusion Criteria: Primary care visit/encounter among people under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500000 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Suicide Risk Safety Plan Documentation | Rates for primary care encounters will be compared before and after implementation, during the 13 month study period 3/05/2025-4/05/2026 (implementation launch 10/6/2025)
  Indicator for whether a patient was identified at risk of suicide (using the PHQ-9 and C-SSRS) and had a safety planning intervention documented in the EMR on the day of, or in the following 14 days of a primary care encounter, using a standardized template based on the brief suicide risk safety plan intervention developed by Drs. Stanley & Brown to mitigate risk

SECONDARY OUTCOMES:
Suicidal ideation symptom assessment | Rates of assessment for primary care encounters will be compared before and after implementation, during the 13 month study period 3/05/2025-4/05/2026 (implementation launch 10/6/2025)
  Indicator for whether a patient completed the Patient Health Questionnaire-9 (PHQ-9) Question 9 for primary care encounter
Prior month intent/planning for suicide attempt | Rates for primary care encounters will be compared before and after implementation, during the 13 month study period 3/05/2025-4/05/2026 (implementation launch 10/6/2025)
  Indicator for whether a patient indicated prior-month intent or planning for suicide attempt (C-SSRS score ≥3, on the C-SSRS assessment for the primary care encounter (range 0-6; higher scores confer greater risk)
Suicide risk assessment | Rates for primary care encounters will be compared before and after implementation, during the 13 month study period 3/05/2025-4/05/2026 (implementation launch 10/6/2025)
  Indicator for whether a patient completed the Columbia Suicide Risk Severity Rating Scale (C-SSRS) for the primary care encounter
Frequent suicidal ideation reported (in prior 2-weeks) | Rates for primary care encounters will be compared before and after implementation, during the 13 month study period 3/05/2025-4/05/2026 (implementation launch 10/6/2025)
  Indicator for whether a patient reported suicidal ideation "more than half the days" or "nearly every day" (PHQ-9 Q9 score 2 or 3), on the assessment documented in the electronic medical record (EMR) for the primary care encounter (range 0-3, higher scores indicate more frequent suicidal ideation)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No